CLINICAL TRIAL: NCT04822545
Title: Inpatient Referral to Comprehensive Weight Management for Patients With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIM-2020-29448
Record Dates: First submitted 2020-12-22; First posted 2021-03-30 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Other): -Adult (≥ 18 years of age) hospitalized patients who have obesity (BMI ≥ 30 kg/m2 or BMI ≥ 27 kg/m2 if Asian/South Asian), as recorded in the medical chart, who have decision-making capacity and whose acute medical condition has been stabilized.
  we will exclude patients who are enrolling in hospice/comfort care and the patients who are already enrolled in the CWM clinic. Non-English speaking patients. Patients who have opted out of research in their Epic EHR will be excluded from consideration for participation.
  Interventions: Other: referral to comprehensive weight management clinic

INTERVENTIONS:
Other: referral to comprehensive weight management clinic — Patients will receive a referral for outpatient CWM clinic, with a message sent to the CWM clinic scheduler, prior to hospital discharge.
  At six months after discharge, the patient will receive a phone call from the investigators to ascertain whether they were able to go to the CWM clinic and about their experience.

SUMMARY:
Hospitalized patients with obesity who are not already in CWM (comprehensive weight management), or not comfort care/hospice will be identified by the hospitalists then the study dietitian will consent for the patient for enrollment (and answer any question regarding diet/lifestyle) in the study. The intervention will be a CWM referral at discharge. The outcome will be what percentage of these patients go to the CWM clinic at 6 months. At 6 months, the investigators will also call each participant to get a qualitative idea of the process of inpatient referral and barriers to the CWM clinic visit. Weight loss, starting on anti-obesity medication, bariatric surgery will be assessed as a secondary outcome.

DETAILED DESCRIPTION:
* The investigators will conduct an uncontrolled, one arm interventional study on Adult (≥ 18 years of age) hospitalized patients who have obesity (BMI ≥ 30 kg/m 2 or BMI ≥ 27 kg/m 2 if Asian/South Asian), and after stabilization of their acute medical conditions. Prior to hospital discharge, patients will receive a referral for an outpatient comprehensive weight management clinic, with a message that will be sent to the CWM clinic scheduler. Then the investigators will follow the patients forward for 6 months from hospital discharge to assess primary and secondary outcomes. Also, the investigators will look at a historical control group of hospitalized patients with obesity (age, comorbidity matched) from 2014-2019 (chosen instead of 2020, to avoid any impact of 2020 COVID 19 pandemic) and compare the primary and secondary outcomes. At six months after discharge, patients will receive a phone call from the investigators to ascertain whether they were able to go to the comprehensive weight management clinic and about their experience.
* Hospitalized patients who have decision-making capacity and whose acute medical condition has been stabilized who meet study criteria will be identified by study physician(s) who will look at his/her personal patient list on a regular basis to identify patients who meet enrollment criteria and will refer the patients to the co-investigator who is not directly involved in the patient's care who will then discuss enrollment with patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age) hospitalized patients who have obesity (BMI ≥ 30 kg/m2 or BMI ≥ 25 kg/m2 if Asian/South Asian)
* Who have decision-making capacity
* Whose acute medical condition has been stabilized.

Exclusion Criteria:

* Patients in the ICU or requiring > 6 LPM of supplemental oxygen
* Patients enrolling in hospice/comfort care
* Patients who are already enrolled in weight management or have undergone previous metabolic / bariatric surgery.
* Non-English speaking patients.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Perform a feasibility study of providing referral to outpatient comprehensive weight management clinic to Inpatients with obesity. | Six months
  Percentage of patients who are seen in weight management clinic at 6 months from hospital discharge

SECONDARY OUTCOMES:
The number of Comprehensive weight managment clinic visits at 6 months. | six month and 12 month
Weight loss at 6 months from hospital discharge. | six month and 12 month
Qualitative information about the experience of getting referral for outpatient weight management while inpatient and experience of going to weight management | six month and 12 month
  Obtained by survey and phone call
Percentage of patients receiving weight-loss medications or being referred for bariatric surgery. | six month and 12 month
Compare primary and secondary outcomes with a historical control of patients with obesity | six month and 12 month
  Historical control will be defined as inpatients with obesity admitted to the same hospital from 2014 to 2019

CONTACTS AND LOCATIONS:
Overall Officials: Nirjhar Dutta, DO, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No